CLINICAL TRIAL: NCT00937677
Title: Effect of Natalizumab (Tysabri®) on Remyelination in Patients With Relapsing-remitting Multiple Sclerosis. A Follow-up Voxel-wise Magnetization Transfer Imaging Study.
Brief Title: Effect of Tysabri in Patients With Relapsing-Remitting Multiple Sclerosis: A Follow-up Magnetization Transfer Imaging (MTI) Study
Status: Completed | Type: Observational
Sponsor: University at Buffalo (Other)
Collaborators: Biogen (Industry)
Responsible Party: Principal Investigator, Robert Zivadinov, MD, PhD, Professor of Neurology, University at Buffalo
Other Study IDs: BNAC/Tysabri/01
Record Dates: First submitted 2009-07-09; First posted 2009-07-13 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2011-09

CONDITIONS: Multiple Sclerosis
Keywords: Tysabri; VWMTR
MeSH Terms: conditions — Multiple Sclerosis | interventions — Natalizumab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: 63 patients with relapsing-remitting Multiple Sclerosis who are enrolled in the TOUCH program and have been taking Tysabri monotherapy for 2 years.
  Interventions: Drug: Tysabri
- 2: 22 age- and sex-matched normal controls who completed 1 year follow-up.

INTERVENTIONS:
Drug: Tysabri — Infusion of TYSABRI® 300 mg in 100 mL 0.9% Sodium Chloride Injection, USP over approximately one hour at month 0 and 12 and 24 months. After the infusion is complete, flush with 0.9% Sodium Chloride Injection, USP.
  Use of filtration devices during administration has not been evaluated. Other medications should not be injected into infusion set side ports or mixed with TYSABRI®.
  TYSABRI® concentrate is supplied as 300 mg natalizumab in a sterile, single-use vial free of preservatives. Each package contains a single-use vial.
  Other Names: Natalizumab
  Groups: 1

SUMMARY:
The primary objective of this study is to define the effect of Tysabri in patients with relapsing-remitting (RR) multiple sclerosis (MS) over 2 years. The investigators will also explore the extent of remyelination in MS patients treated with Tysabri over 2 years.

A secondary objective of this study is to investigate differences in the capacity for remyelination between patients who do or do not respond to Tysabri monotherapy during the same 24 months.

A tertiary objective of this study is to monitor Tysabri effect in MS antiphospholipid antibodies positive and MS antiphospholipid antibodies negative patients and to determine perfusion differences according to the antiphospholipid antibodies positivity status.

DETAILED DESCRIPTION:
Magnetization transfer imaging (MTI) is a widely used tool for characterizing the evolution of multiple sclerosis (MS) lesions and normal appearing brain tissue (NABT). As remyelination and demyelination are heterogeneous in each lesion and NABT, techniques such as voxel-wise based MTR dynamic mapping may help predict an individual's clinical course, as well as the effect of treatment, by revealing evidence of myelin repair and neuroprotection.

Natalizumab (Tysabri) showed a robust effect on the decrease of inflammation in phase II and III clinical trials, as evidenced by the decrease in Gd enhancing and T2 lesions and on the decrease of clinical activity as measured by reduction of clinical relapses and progression of disability. The effect of Tysabri on non-conventional measures is only partially known.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with clinically definite MS according to the Polman criteria
* Age 18-65
* Have a RR disease course
* Have EDSS scores less than or equal to 5.5 {Kurtzke, 1983 #15}
* Have disease duration less than 20 years
* Fulfilled the TOUCH enrollment requirements and started on Tysabri monotherapy
* Signed informed consent
* None of the exclusion criteria

Exclusion Criteria:

* Primary progressive, secondary progressive, or progressive relapsing MS. Primary progressive, secondary progressive or progressive relapsing multiple sclerosis.
* A clinically significant infectious illness (e.g., cellulitis, abscess, pneumonia, septicemia) within 30 days prior to drug start.
* History of, or abnormal laboratory results indicative of, any significant cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, gastrointestinal, dermatologic, psychiatric, renal, and/or other major disease that, in the opinion of the investigator, would preclude the administration of natalizumab for the duration of the study.
* History of severe allergic or anaphylactic reactions or known drug hypersensitivity.
* Abnormal blood tests, performed at the screening visit, which exceed any of the limits defined below:
* ALT/ SGPT, or AST/ SGOT > three times the upper limit of normal (i.e., 3xULN).
* Total white blood cell (WBC) count <2,300/mm3.
* Platelet count <100,000/mm3.
* Creatinine > 2xULN.
* Prothrombin time (PT) > ULN.
* Any prior treatment during the 2 weeks prior to study screening with agents such as IFN-β, GA, IVIG, or on the following immunosuppressant therapies for less than 3 months: mitoxantrone, cyclophosphamide, cladribine, fludarabine, cyclosporine, azathioprine, methotrexate, Cellcept, etc.
* History of alcohol or drug abuse within 2 years prior to randomization.
* Female subjects who are not postmenopausal for at least 1 year, surgically sterile, or willing to practice effective contraception (as defined by the investigator) during the study. The rhythm method is not to be used as the sole method of contraception.
* Nursing mothers, pregnant women, and women planning to become pregnant while on study.
* Unwillingness or inability to comply with the requirements of this protocol including the presence of any condition (physical, mental, or social) that is likely to affect the subject's ability to comply with the study protocol.
* Any other reasons that, in the opinion of the Investigator, indicate that the subject is unsuitable for enrollment into this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: MS patients that are followed at the Jacobs Neurological Institute, University at Buffalo, Buffalo NY.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2007-11; Primary Completion 2009-12 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
To define the effect of Tysabri monotherapy on a voxel-wise basis using magnetization transfer ratio dynamic mapping of the lesions and normal appearing brain tissue in patients with relapsing-remitting multiple sclerosis. | 2 years

SECONDARY OUTCOMES:
To investigate differences in the capacity for remyelination measured by MTR between patients who do or do not respond to Tysabri monotherapy. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Robert Zivadinov, MD, PHd, Principal Investigator — University at Buffalo
Locations (1):
- Jacobs Neurological Institute, Buffalo, New York, United States

REFERENCES:
- [Derived] Zivadinov R, Dwyer MG, Hussein S, Carl E, Kennedy C, Andrews M, Hojnacki D, Heininen-Brown M, Willis L, Cherneva M, Bergsland N, Weinstock-Guttman B. Voxel-wise magnetization transfer imaging study of effects of natalizumab and IFNbeta-1a in multiple sclerosis. Mult Scler. 2012 Aug;18(8):1125-34. doi: 10.1177/1352458511433304. Epub 2011 Dec 22. PMID 22194217